CLINICAL TRIAL: NCT03873155
Title: The Effectiveness of Mindfulness Based Cognitive Group Therapy for Social Anxiety Symptoms in People Living With Alopecia Areata: A Single Group Case Series.
Brief Title: The Effectiveness of Mindfulness Based Cognitive Group Therapy for Social Anxiety Symptoms in People Living With Alopecia Areata
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sheffield (Other)
Collaborators: Alopecia UK (Unknown)
Responsible Party: Principal Investigator, Andrew Thompson, Principal Investigator, University of Sheffield
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 230374
Record Dates: First submitted 2019-03-04; First posted 2019-03-13 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Alopecia Areata; Social Anxiety
MeSH Terms: conditions — Alopecia Areata | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Intervention Model Description: A single-group case-series design will be adopted, whereby one group of participants will complete daily and weekly measures over the course of 1) a 4-week randomised multi-baseline period; 2) a 9-week intervention period (one introductory week added on to usual structure); 3) a 4-week follow up-period. Variables collected during the intervention and follow-up period will be compared with those from the baseline period.
Masking Description: No party will be masked in this study. There is only one arm and participants will act as their own controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness-based cognitive therapy (Experimental): There is only one arm in this study. A range of variables will first be measured (daily and weekly) over a baseline period in a group of participants. Following this baseline period, participants will be take part in an MBCT intervention whilst the same variables are measured. Following the intervention,there will be a 4-week follow-up period, and MBCT groups will not run during this time.
  Interventions: Behavioral: Mindfulness Based Cognitive Therapy

INTERVENTIONS:
Behavioral: Mindfulness Based Cognitive Therapy — Mindfulness based cognitive group therapy (MBCT) is a structured eight-week programme (although an extra introductory week will be added in the current study) that combines mindfulness-based exercises with cognitive therapy.

SUMMARY:
This study investigates the impact of mindfulness based cognitive therapy (MBCT) on social anxiety in adults with alopecia areata. A single-group case-series design will be adopted.

DETAILED DESCRIPTION:
Alopecia areata (AA) is an immunological disorder which is characterised by round/oval patches of non-scarring hair loss. People living with AA are at higher risk of developing depression, anxiety and social phobia than the general population (Koo et al., 1994; Ruiz-Doblado, Carrizosa, & García-Hernández, 2003). Interventions that aim to reduce engagement in negative appearance related thoughts, and attentional bias towards negative self-referential information may be helpful for this population.

Mindfulness-based cognitive therapy (MBCT) offers one potential method of reducing social anxiety in individuals with AA. MBC is a structured eight-week programme that has been recommended by the National Institute of Clinical Excellence as an effective intervention to reduce the risk of relapse in depression since 2009.

The main aim of the current study is to investigate whether an MBCT course can reduce social anxiety in individuals with AA. A single-group case-series design will be adopted, whereby participants will act as their own control; data collected from participants during and after they have received the intervention will be compared to data collected before they have received the intervention. Semi-structured interviews will be carried out at the end of the study to investigate participants experiences of the intervention.

The investigators predict that MBCT will reduce social anxiety in individuals with AA. More specifically, the hypothesis are:

(i) participants will experience an increase in mindfulness during the intervention period, relative to the baseline phase and this will be maintained at follow-up

(ii) increases in mindfulness will be associated with decreases in social anxiety, anxiety and depression, and increases in dermatology quality of life.

ELIGIBILITY:
Inclusion Criteria:

* AA is the main presenting physical health problem
* Participant self-identifies as experiencing social anxiety
* Sufficient English to participate in group sessions and discussion.
* Aged 16 and over

Exclusion Criteria:

* Primary psychiatric diagnosis affecting skin (e.g., trichotillomania)
* Hair loss as a result of medical intervention or surgery (e.g., chemotherapy)
* The skin condition is secondary to other physical health problems (e.g., arthritis, cancer, chronic pain)
* Patient does not report any social distress as a result of their AA
* Currently undergoing other psychological therapy

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-09-23 (Actual)

PRIMARY OUTCOMES:
Change in social anxiety (idiosyncratic measure) | Daily for 20 weeks (baseline-intervention-follow-up)
  The primary outcome measures for the proposed study are idiosyncratic measures of social anxiety which will be assessed daily by text message. Participants will be asked to identify one social anxiety-related positive target (something the participant would like to improve) and one negative target (something the participant would like to reduce). Participants will respond to the daily text messages with a score on a 0-100 scale

SECONDARY OUTCOMES:
Social Anxiety | Weekly for 21 weeks (baseline-intervention-follow-up)
  The Brief Fear of Negative Evaluation straight forward items (BFNE-S: Carleton, Collimore, McCabe, & Antony, 2011) will be used to assess social anxiety. The measure consists of 8 questions rated on a 5-point Likert scale (from "not at all characteristic of me" to "entirely characteristic of me").
Mindfulness | Weekly for 21 weeks (baseline-intervention-follow-up)
  The Five Factor Mindfulness Questionnaire-15 (FFMQ-15; Baer, Carmody, & Hunsinger, 2012) will be used to measure mindfulness. Items are rated on a five-point Likert scale (from "never or very rarely true" to "very often or always true").
Mindfulness | 4 time-points. Assessment (beginning of study) beginning of intervention (4 weeks later) end of intervention (9 weeks later) follow-up (8 weeks later)
  The Five Factor Mindfulness Questionnaire (FFMQ; Baer, Smith, Hopkins, Krietemeyer & Toney, 2006) will also be used to measure mindfulness. Items are rated on a five-point Likert scale (from "never or very rarely true" to "very often or always true").
Depression | 4 time-points. Assessment (beginning of study) beginning of intervention (4 weeks later) end of intervention (9 weeks later) follow-up (8 weeks later)
  The 9-item self-report Patient Health Questionnaire (PHQ-9; Spitzer, Kroenke, & Williams, 1999) will be used to measure symptoms of depression. Items are rated on a four-point Likert scale (from "not at all" to "nearly every day").
Anxiety | 4 time-points. Assessment (beginning of study) beginning of intervention (4 weeks later) end of intervention (9 weeks later) follow-up (8 weeks later)
  The Generalised Anxiety Disorder Questionnaire (GAD-7; Spitzer, Kronke, Williams, & Lowe, 2006) is a 7 item self-report scale to measure generalized anxiety symptoms. Items are rated on a four-point Likert scale (from "not at all" to "nearly every day").
Quality of life (dermatology-related) | 4 time-points. Assessment (beginning of study) beginning of intervention (4 weeks later) end of intervention (9 weeks later) follow-up (8 weeks later)
  The Dermatology Quality of Life Index (DLQI: Findlay & Khan, 1994) consists of 10 questions concerning the impact of the skin condition over the last week. Questions relate to symptoms and feelings, daily activity, leisure, work/school, personal relationships and side effects of treatment. Items are rated on a 4-point Likert scale (from "not at all" to "very much").
Service use | 3-time points. 4 time-points. Beginning of intervention (4 weeks after assessment) end of intervention (9 weeks later) follow-up (8 weeks later)
  The Client Service and Receipt Inventory (CSRI; Beecham & Knapp, 2001) is a 6 question measure of client service utilization. More specifically, the CSRI measures how often participants have met with a healthcare professional, visited A & E, been an inpatient, used an ambulance, received a diagnostic test, and days spent away from work due to ill health.
Work and social adjustment | 3-time points. 4 time-points. Beginning of intervention (4 weeks after assessment) end of intervention (9 weeks later) follow-up (8 weeks later)
  The Work and Social Adjustment Scale (WSAS; Mundt & Marks, 2002) is a 5-item measure of the impact of mental health issues on an individual's social life and ability to work.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - The University of Sheffield, Sheffield, South Yorkshire
  - Royal Hallamshire Hospital (Sheffield Teaching Hospital), Sheffield, South Yorkshire

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Koo JY, Shellow WV, Hallman CP, Edwards JE. Alopecia areata and increased prevalence of psychiatric disorders. Int J Dermatol. 1994 Dec;33(12):849-50. doi: 10.1111/j.1365-4362.1994.tb01018.x. PMID 7883407
- [Background] Ruiz-Doblado S, Carrizosa A, Garcia-Hernandez MJ. Alopecia areata: psychiatric comorbidity and adjustment to illness. Int J Dermatol. 2003 Jun;42(6):434-7. doi: 10.1046/j.1365-4362.2003.01340.x. PMID 12786868
- [Background] Carleton RN, Collimore KC, McCabe RE, Antony MM. Addressing revisions to the Brief Fear of Negative Evaluation scale: measuring fear of negative evaluation across anxiety and mood disorders. J Anxiety Disord. 2011 Aug;25(6):822-8. doi: 10.1016/j.janxdis.2011.04.002. Epub 2011 Apr 16. PMID 21565463
- [Background] Baer RA, Carmody J, Hunsinger M. Weekly change in mindfulness and perceived stress in a mindfulness-based stress reduction program. J Clin Psychol. 2012 Jul;68(7):755-65. doi: 10.1002/jclp.21865. Epub 2012 May 23. PMID 22623334
- [Background] Baer RA, Smith GT, Hopkins J, Krietemeyer J, Toney L. Using self-report assessment methods to explore facets of mindfulness. Assessment. 2006 Mar;13(1):27-45. doi: 10.1177/1073191105283504. PMID 16443717
- [Background] Spitzer RL, Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. Primary Care Evaluation of Mental Disorders. Patient Health Questionnaire. JAMA. 1999 Nov 10;282(18):1737-44. doi: 10.1001/jama.282.18.1737. PMID 10568646
- [Background] Finlay AY, Khan GK. Dermatology Life Quality Index (DLQI)--a simple practical measure for routine clinical use. Clin Exp Dermatol. 1994 May;19(3):210-6. doi: 10.1111/j.1365-2230.1994.tb01167.x. PMID 8033378
- [Background] Beecham, J. and Knapp, M. (2001) Costing psychiatric interventions, in G. Thornicroft (ed.) Measuring Mental Health Needs, Gaskell, 2nd edition, 200-224.
- [Background] Mundt JC, Marks IM, Shear MK, Greist JH. The Work and Social Adjustment Scale: a simple measure of impairment in functioning. Br J Psychiatry. 2002 May;180:461-4. doi: 10.1192/bjp.180.5.461. PMID 11983645